CLINICAL TRIAL: NCT05379491
Title: An Efficacy and Safety Evaluation of Linaclotide in Bowel Preparation by Patients at High Risk of Inadequate Bowel Preparation: a Multicenter, Randomized, Double-Blind, Controlled Clinical Trial
Brief Title: Application of Linaclotide Capsule in Bowel Preparation for Patients at High Risk of Inadequate Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhiguo Liu (Other)
Responsible Party: Sponsor-Investigator, Zhiguo Liu, Associate Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KY20222119-F-1
Record Dates: First submitted 2022-05-14; First posted 2022-05-18 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Colonoscopy
Keywords: colonoscopy; inadequate bowel preparation; Boston Bowel Preparation Scale; linaclotide
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomized grouping sequence by block randomization with a block size of 4 is generated using a web-based service. Linaclotide or placebo is allocated according to the sequence and labelled in numerial order (1 - 720) without labelling the allocation information. Therefore, patients, endoscopists, and other investigators at each center will be unaware of the drug allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 L PEG + Linaclotide (Active Comparator): Bowel preparation for colonoscopy was performed with 3 L polyethylene glycol solution combined with 2-day linaclotide.
  Interventions: Drug: 3 L PEG + linaclotide
- 3 L PEG + Placebo (Placebo Comparator): Bowel preparation for colonoscopy was performed with 3 L polyethylene glycol solution combined with 2-day placebo.
  Interventions: Drug: 3 L PEG + placebo

INTERVENTIONS:
Drug: 3 L PEG + linaclotide — Participants take a linaclotide capsule on the day before colonoscopy at least 30 minutes before the first meal (if this is impossible, take the capsule as early as possible on that day). Participants take 1 L polyethylene glycol electrolyte solution within 1 hour from 8 p.m the night before the examination and take another linaclotide capsule and 2 L polyethylene glycol electrolyte solution 4 hours before the colonoscopy.
  Arms: 3 L PEG + Linaclotide
Drug: 3 L PEG + placebo — Participants take a placebo capsule on the day before colonoscopy at least 30 minutes before the first meal (if this is impossible, take the capsule as early as possible on that day). Participants take 1 L polyethylene glycol electrolyte solution within 1 hour from 8 p.m the night before the examination and take another placebo capsule and 2 L polyethylene glycol electrolyte solution 4 hours before the colonoscopy.
  Arms: 3 L PEG + Placebo

SUMMARY:
The purpose of this study is to compare the colon cleansing quality of linaclotide versus control in adult patients at high risk of inadequate bowel preparation: one group will receive polyethylene glycol solution (PEG) split dose (1 L + 2 L) plus linaclotide and the other group PEG (1 L + 2 L) plus placebo before colonoscopy.

DETAILED DESCRIPTION:
The objective of this trial is to compare the colon cleanliness achieved with PEG split dose (1 L + 2 L) + linaclotide versus PEG split dose (1 L + 2 L) + placebo for patients scheduled for a colonoscopy at high risk of inadequate bowel preparation. The target patients are those with constipation, poor bowel preparation history, history of abdominal/pelvic surgery, comorbidity (diabetes, Parkinson's disease, stroke, or history of spinal cord injury), BMI > 25 kg/m2, age > 70, tricyclic antidepressants usage, or opioid usage, as defined by the latest version of Bowel Preparation Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for colonoscopy
* age ≥ 18
* meet any of the followings: functional constipation according to Rome IV criteria, poor bowel preparation history, BMI > 25 kg/m2, age > 70, history of abdominal/pelvic surgery, comorbidity (diabetes, Parkinson's disease, stroke, or history of spinal cord injury), antidepressant usage, opioid usage
* willing to provide informed consent

Exclusion Criteria:

* unable to cooperate with questionnaires
* uncontrolled hypertension (systolic .170 mm Hg and diastolic.100mmHg)
* pregnancy or lactation
* toxic colitis, or megacolon
* allergy to preparation components
* active inflammatory bowel disease
* clinically significant electrolyte abnormalities
* a history of severe renal, liver, or cardiac insufficiency
* has already been enrolled in the study
* gastrointestinal obstruction
* obvious gastroparesis or gastric retention
* bowel perforation
* polyp syndrome
* history of colectomy
* any other condition that is inappropriate for enrollment as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Bowel preparation adequate rate | 48 hours
  The rate of participants with all colon segment scores (proximal colon, transverse colon, distal colon) are ≥ 2 according to Boston Bowel Preparation Scale.
Number of adenomas per patient | 48 hours
  If there is no significant difference in the first primary outcome between the two groups, compare the average number of adenomas per patient detected by colonoscopy.

SECONDARY OUTCOMES:
Subject willingness to repeat the preparation | 1 Day of colonoscopy
  Survey
Tolerance to bowel preparation | 1 Day of colonoscopy
  It will be subjective and assessed as non, mild, moderate, severe.
Tolerance to colonoscopy | 1 Day of colonoscopy
  It will be subjective and assessed as non, mild, moderate, severe.
Average number of polyps per patient | 1 Day of colonoscopy
  Average number of polyps detected per patient by colonoscopy in each arm
Average number of adenomas per patient | 1 Day of colonoscopy
  Average number of adenomas detected per patient by colonoscopy in each arm
Withdrawal time | 1Day of colonoscopy
  the time from cecal identification to the withdrawal of the colonoscopy across the anus minus the time of polypectomy.
Cecal intubation rate for colonoscopies | 1 Day of colonoscopy
  Cecal intubation was defined as reaching the ileocecal valve

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, M.D., Principal Investigator — Study Principal Investigator
Locations (8):
- China (8):
  - Ningxia Hui Autonomous Region People's Hospital, Yinchuan, Ningxia
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Xi'an Jiaotong University Second Affiliated Hospital, Xi'an, Shaanxi
  - Air Force 986 Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No